CLINICAL TRIAL: NCT01528501
Title: An Open-label, Uncontrolled Phase II Trial of HDAC-Inhibitor LBH589 in Patients With Chemo-refractory Metastatic Gastric Cancer Overexpressing Histone Deacetylases (HDACs) - CLBH589BDE03T
Brief Title: Histone Deacetylases - Gastric Cancer (HDAC-GaCa-2008)
Acronym: HDAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: medical/ethical reasons
Sponsor: Technical University of Munich (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BDE03T
Record Dates: First submitted 2012-02-01; First posted 2012-02-08 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Panobinostat

ARMS (1):
- I (Experimental)
  Interventions: Drug: Panobinostat (LBH589)

INTERVENTIONS:
Drug: Panobinostat (LBH589)

SUMMARY:
This is an open-label, phase II trial evaluating the antitumor activity and safety of the oral Histone Deacetylase (HDAC)-Inhibitor LBH589. The treatment consists of 20 mg LBH589 three times a week in patients with chemo-refractory HDAC overexpressing.

metastatic adenocarcinoma of stomach, esophagogastric junction or lower esophagus (Barrett carcinoma). One cycle lasts 21 days. A total of 28 patients will be enrolled in this trial. In patients experiencing LBH589-related toxicity requiring treatment rest or dose reduction dose may be reduced. Subsequent dose adjustment will be permitted based on outcome. Treatment will continue until disease progression or intolerable adverse events. Subsequently, the patients will be followed-up for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 - 90 years
2. Signed and dated informed consent of the patient before the start of specific protocol procedures
3. Histologically proven adenocarcinoma of stomach, esophagogastric junction or lower esophagus (Barrett carcinoma)
4. Measurable metastatic disease according to the RECIST (33). If locally recurrent disease, it must be associated with at least one measurable lymph node (> 20 mm by CT scan or > 10 mm with spiral CT)
5. Overexpression of at least one class I HDAC in the cancer biopsy as assessed by immunohistochemistry
6. Failure of prior palliative chemotherapy/chemotherapies (at least one Irinotecan- or Cisplatin-based). Failure is defined either by progression of disease or by significant toxicity that precludes further treatment
7. At least 4 weeks from previous chemotherapy at first dose of trial drug
8. Resolution of all acute toxic side effects of prior therapy or surgical procedures to grade ≤ 1 NCI-CTC (except for the laboratory values)
9. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤ 1.5 x ULN
   * Absolute neutrophil count (ANC) ≥ 1500/µL
   * Platelets ≥ 100,000/µL
   * Hemoglobin ≥ 8.0 g/dL without support of growth factors (previous administration of erythrocyte concentrate is allowed)
   * Calculated CrCl ≥ 50 mL/min (MDRD Formula)
   * Serum calcium ≤ 12.0 mg/dL
   * Serum creatinine ≤ 2.0 x ULN
   * Lipase/Amylase ≤ 2,5 x ULN
   * All other laboratory values specified in chapter 7.5: resolution of all side effects of prior therapy or surgical procedure to grade < 3 NCI CTC
10. At least 4 weeks from any major surgery (at first dose of trial drug)
11. Karnofsky Performance Status (KPS) > 70
12. Life expectancy > 12 weeks
13. Patients must be able to swallow LBH589 capsules
14. Patients who understand the nature of the trial and are willing and able to comply with scheduled visits, treatment plans, laboratory tests and other trial procedures
15. Female patients who are capable of bearing children must have a negative pregnancy test result (serum or urine) at trial entry. All women included in the trial must be surgically sterile or postmenopausal or agree to employ adequate birth control measures for the duration of the trial and six months post-dosing. Male patients must be surgically sterile or must agree to use effective contraception during the trial and six months post-dosing

Exclusion Criteria:

1. Other tumor type than adenocarcinoma (e.g., leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix which has been effectively treated. Patients curatively treated and disease free for at least 5 years will be discussed with the sponsor before inclusion
2. Patients with known brain or leptomeningeal metastasis
3. Intake of non-permitted concomitant drugs (the coordinating investigator should be contacted to discuss the individual case), see chapter 5.4:

   * Concomitant treatment with antiarrhythmics and drugs with dysrhythmic potential (ie, terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, and indapamide)
   * Prior exposure to a HDAC inhibitor compound
   * Administration of potent CYP34A inhibitors during or within 7 days before start of LBH589-treatment (e.g. ketoconazole, itraconazole, clarithromycin, erythromycin, diltiazem, verapamil, delavirdine, indinavir, saquinavir, ritonavir, atazanavir, nelfinavir, grapefruit juice)
   * Administration of potent CYP3A4 inducers during or within 12 days before start of LBH589-treatment (e.g. dexamethasone, rifampicin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John´s wort, efavirenz, tipranavir)
   * Ongoing treatment with therapeutic doses of anticoagulants such as Coumadin or heparins (however, low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed)
   * Any other medicinal anticancer therapy during treatment phase except treatment with non-conventional therapies (e.g. herbs or acupuncture) and vitamins/mineral supplements, provided that they do not interfere with the trial endpoint, in the opinion of the investigator
   * Concurrent systemic immune therapy, chemo- or hormone therapy
   * Concomitant or within a 4-week period administration (from first dose of trial drug) of any other experimental drug under investigation) and participation in another clinical trial
4. Any prior radiotherapy of target lesions
5. Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (> hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis
6. Current history of chronic diarrhea and/or diarrhea > CTCAE grade 3
7. Active disseminated intravascular coagulation, or patients prone to thromboembolism
8. Known human immunodeficiency virus (HIV) infection
9. Active uncontrolled infection
10. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with trial participation or trial drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into the trial
11. Known allergic/hypersensitivity reaction to any of the components of the treatment; or known drug abuse/alcohol abuse
12. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

    * Known history of QT interval prolongation, ongoing QT prolongation (> 450 msec for males or > 470 msec for females), any cardiac ventricular dysrhythmias, atrial fibrillation of any grade
    * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with the Sponsor prior to enrollment)
    * Any history of ventricular fibrillation or torsade de pointes
    * Bradycardia defined as HR < 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
    * Screening ECG with a QTc > 450 msec
    * Right bundle branch block + left anterior hemiblock (bifascicular block)
    * Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
    * Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
13. Patients who have received steroids (e.g. dexamethasone) ≤ 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy. Concomitant therapy medications that include corticosteroids are allowed if patients receive < 10 mg of prednisone or equivalent as indicated for other medical conditions, or up to 100 mg of hydrocortisone as pre-medication for administration of certain medications or blood products while enrolled in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
objective response rate within the first six treatment cycles
  objective response rate (CR + PR) within the first six treatment cycles

SECONDARY OUTCOMES:
Progression free survival (PFS)
1-year survival
Overall survival
Safety and tolerability of LBH 589
  Analysis of adverse events and laboratory data

CONTACTS AND LOCATIONS:
Overall Officials: Martina Mayr, Dr., Principal Investigator — Klinikum rechts der Isar
Locations (2):
- Germany (2):
  - Klinikum rechts der Isar, Munich, Bavaria
  - Universitätsklinikum Mannheim, Mannheim